CLINICAL TRIAL: NCT03025503
Title: Nipple Stimulation for Labor Induction: Efficiency, Safety and Satisfaction Measures
Brief Title: Nipple Stimulation for Labor Induction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NippleStim-HMO-CTIL
Record Dates: First submitted 2016-12-18; First posted 2017-01-19 (Estimated); Last update posted 2017-01-19 (Estimated); Status verified 2016-12

CONDITIONS: Delivery Delayed

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- nipple stimulation (Experimental)
  Interventions: Other: nipple stimulation
- no intervention (No Intervention)

INTERVENTIONS:
Other: nipple stimulation
  Arms: nipple stimulation

SUMMARY:
This study will examine the use of nipple stimulation for cervical ripening in women who present to the labor and delivery ward after their water has broken but have a contraindication to prostaglandins.

ELIGIBILITY:
Inclusion Criteria:

* Week 37 + 0 and on
* PROM (premature rupture of membranes)
* Multiparity (birth sixth or higher) or TOLAC (trial of labor after Caesarean section)
* Not in active labor - without regular contractions fetal monitor, cervical dilation < 4 cm and effacement < 80%.

Exclusion Criteria:

* Water break > 24 hours at the time of admission to the delivery room
* Active vaginal bleeding with suspected placental abruption
* Maternal fever
* Multifetal pregnancy
* Women with contraindication for vaginal birth
* Preeclampsia
* IUGR (intrauterine growth restriction)
* Macrosomia
* Non-reassuring fetal heart tracing

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-01; Primary Completion 2018-01 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
progression to active labor as measured by the Bishop score | 6 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: Undecided